CLINICAL TRIAL: NCT00064051
Title: A Phase II Study of Triapine in Combination With Gemcitabine in Patients With Pancreatic Cancer
Brief Title: 3-AP and Gemcitabine in Treating Patients With Unresectable or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: VION-CLI-031; CDR0000306461 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-08

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine use different ways to stop tumor cells from dividing so they stop growing or die. 3-AP may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth and may help gemcitabine kill more cancer cells by making them more sensitive to the drug.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with 3-AP works in treating patients with unresectable or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate (partial and complete response) in patients with unresectable or metastatic pancreatic cancer treated with 3-AP and gemcitabine.
* Determine the progression-free interval and survival of patients treated with this regimen.
* Determine the safety and feasibility of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Stage I: Patients receive 3-AP IV over 4 hours and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
* Stage II: Patients receive a higher dose of 3-AP IV continuously over 24 hours on days 1, 8, and 15. Within 1 hour of completing 3-AP administration, patients receive gemcitabine IV over 30 minutes on days 2, 9, and 16. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month, every 2 months for 6 months, and then every 3 months for 18 months.

PROJECTED ACCRUAL: A total of 50-95 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic cancer

  * Unresectable or metastatic disease
* Measurable disease

  * Outside prior radiation ports OR within prior radiation port if evidence of disease progression after radiotherapy
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* AST and ALT no greater than 3 times upper limit of normal (ULN) (5 times ULN in the presence of liver metastases)
* Chronic viral hepatitis allowed

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 3 months
* No uncontrolled congestive heart failure
* No uncontrolled coronary artery disease
* No uncontrolled arrhythmias

Pulmonary

* No dyspnea at rest
* No dependence on supplemental oxygen

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No other malignancy except any of the following:

  * Carcinoma in situ of the cervix treated with cone biopsy or resection
  * Nonmetastatic basal cell or squamous cell skin cancer
  * Any stage I malignancy curatively resected more than 5 years ago
* No active infection
* No known or suspected glucose-6-phosphate dehydrogenase deficiency
* No other concurrent life threatening illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior vaccines, antibodies, cytokines, or small molecule cell signaling inhibitors allowed

Chemotherapy

* No prior cytotoxic chemotherapy for unresectable or metastatic pancreatic cancer

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* More than 3 weeks since prior surgery and recovered

Other

* More than 3 weeks since prior noncytotoxic treatment regimens and objective evidence of progressive disease
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2006-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate (partial and complete response) as assessed by RECIST criteria

SECONDARY OUTCOMES:
Progression-free and overall survival
Safety and feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (7):
- United States (4):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana Oncology Hematology Consultants, Indianapolis, Indiana
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
- Universitair Ziekenhuis Gent, Ghent, Belgium
- United Kingdom (2):
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England